CLINICAL TRIAL: NCT05212415
Title: Reported Bruxism and Parafunctional Oral Habits in Children and Adolescents With Spastic Cerebral Palsy: a Cross-sectional Study
Brief Title: Bruxism and Parafunctional Oral Habits in Children and Adolescents With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aysenur Tuncer, PT, PhD, Hasan Kalyoncu University
Other Study IDs: 2020/035
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Bruxism
Keywords: Cerebral Palsy; Children; Adolescent; Bruxism; Habits
MeSH Terms: conditions — Cerebral Palsy; Bruxism; Habits

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with CP: Children and adolescents with spastic CP are the group of the observational study.

SUMMARY:
The aim of the study is to evaluate and analyze the rates and relationships between bruxism, other parafunctional oral activities, and oral-motor activities in children and adolescents with spastic CP.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on children and adolescents with CP receiving care services in three different private rehabilitation centers between January 2020 and March 2021. All the parents or primary caregivers included in the study were mothers of children with CP. Initially, information about bruxism and parafunctional oral habits and the study's aims were given to the mothers. All the mothers provided written informed consent for voluntary participation.

63 children and adolescents with spastic CP were analyzed, comprising 35 girls and 28 boys.

All the children were observed in clinical environments for classification according to the Gross Motor Function Classification System (GMFCS) and levels of activity and communication.

Data were collected from an evaluation form, clinical examination of the individuals, and interviews with the mothers.

In the first section of the evaluation, the medical records of the children with CP were reviewed for demographics, and clinical data, including age, gender, CP type, medication, and history of epilepsy. The GMFCS was used to determine the level of impairment in gross motor functions of the children.

In the second section of the evaluation, bruxism and other parafunctional oral activities were evaluated in detail through a face-to-face interview with each child's mother.

Other parafunctional oral habits were both questioned and observed in the clinical environment. The presence of sucking habits (thumb sucking, lip-biting, nail-biting, and cheek biting) and the use of a pacifier for more than 24 months was noted and recorded as present or absent.

The tongue-thrust reflex evaluation scale was applied for tongue thrust. Swallowing problems were evaluated with the water swallowing test, drooling with the saliva control problem severity, and frequency scale.

The habit of chronic breathing through the mouth was evaluated through information gained from the mother and from observation of whether nasal or buccal breaths were taken during routine treatment and evaluation in the clinical environment. For the evaluation of chewing problems, information about feeding was obtained from the mother and recorded as difficulty in chewing solid food, otherwise as absent.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with a diagnosis of spastic CP.
* Children and adolescents ages between 3-18 years old.

Exclusion Criteria:

* Children and adolescents with a diagnosis of dyskinetic, ataxic, and/or mixed type CP
* were aged <3 years or ≥19 years,
* had severe sight or hearing impairment, or had received any orthodontic treatment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The evaluation was made of 63 children and adolescents with spastic CP, comprising 34 (54%) females and 29 (46%) males with a mean age of 9.00±4.26 years.
  The GMFCS level distribution was determined at the highest rate of level 1 in 15 (23.8%) and the lowest level 5 in 9 (14.3%) children.
  Bruxism was present in 33 (52.4%) children, chronic mouth breathing in 33 (55.5%), sucking habits in 21 (33.3%), pacifier use for more than 24 months in 20 (31.7%), and tongue thrust in 13 (20.6%). The results of the oral-motor activity evaluation determined chewing difficulty in 35 (55.5%) children, swallowing problems in 20 (31.7%), and drooling in 23 (36.5%).
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
The GMFCS level | January 2020 and March 2021
  The GMFCS is a widely used, valid, and reliable, standardized system that classifies the impairment of gross motor functions of children with CP in 5 levels (I-II: mild; III: moderate; and IV-V: severe) based on the disabilities and level of dependence.
Parental reported Bruxism | January 2020 and March 2021
  The mothers of the children in the study were given information about bruxism and parafunctional habits. They were then asked, "During the past six months, have you noticed noises of your child clenching or grinding their teeth either when awake or at least three nights a week when sleeping?". The responses were recorded as parental-reported bruxism present or absent.
The Tongue Thrust Rating Scale (TTRS) | January 2020 and March 2021
  The TTRS scale evaluates the tongue's position inside the mouth in four different locations. Tongue position is expressed in figures from 0 to 3, where 0 = none (the tongue is not outside the mouth), 1=mild (tongue between the teeth), 2= moderate (tongue between the lips), and 3= severe (tongue outside the mouth).
Drooling Severity and Frequency Scale | January 2020 and March 2021
  The DSFS, developed by Thomas-Stonell and Greenberg in 1988, is used to determine the level of the saliva control problem. 23 According to the information from the mothers and observation findings, drooling severity was scored from 1-5 and drooling frequency from 1-4. The severity points are interpreted as 1 = no drooling, dry lips, 2=mild, 3= moderate, 4= severe, and 5= excessive drooling wetting the clothes. The frequency points are interpreted as 1=never, 2= occasionally, 3= often, and 4=continuously.
Water Swallowing Test (WST) | January 2020 and March 2021
  In this WST, the subjects in the study were seated and instructed to drink 10 ml of room temperature water. The time taken to drink all the water was recorded. Delayed swallow initiation, drooling, coughing, throat clearing, or a change in voice quality may indicate a problem. After the swallow, the patient should be observed for a minute or more to see a delayed cough response. According to the test evaluation criteria, a score of 1=normal swallowing ability, 2=a likelihood of reduced swallowing ability, and 3= reduced swallowing ability.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PD, Study Director — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided